CLINICAL TRIAL: NCT00796484
Title: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of XL888 in Subjects With Solid Tumors
Brief Title: Safety Study of Pharmacokinetics of XL888 in Adults With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL888-001
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Cancer
Keywords: Cancer; Solid Tumors
MeSH Terms: conditions — Neoplasms

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: XL888

INTERVENTIONS:
Drug: XL888 — Administered orally

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of XL888 in subjects with solid tumors. XL888 is a potent and selective inhibitor of HSP90, a key component of a molecular chaperone complex that promotes the conformational maturation and stabilization of diverse client proteins. Many HSP90 client proteins play critical roles in signaling pathways implicated in tumor cell growth, proliferation, and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a histologically-confirmed tumor that is metastatic or unresectable and is no longer responding to therapies known to prolong survival or to other standard therapies, or has disease for which no effective therapy exists.
2. For subjects enrolling in the maximum tolerated dose expansion cohorts:

   * Subject has documented evidence of Her2-overexpressing tumor; OR
   * Subject has NSCLC that has progressed after a prior response to erlotinib or gefitinib; OR
   * Subject has histologically-confirmed, metastatic melanoma.
   * For subjects in the expansion cohorts A and C: tumor tissue must be accessible for biopsy and subjects must be willing to undergo tumor biopsy.
3. The subject is ≥ 18 years old.
4. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
5. The subject's weight is ≥ 40 kg.
6. The subject has adequate organ and marrow function.
7. The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.
8. Sexually active subjects (male and female) must use accepted methods of contraception during the course of the study and for 3 months after the last dose of XL888.
9. Female subjects of childbearing potential must have a negative pregnancy test at screening.

Exclusion Criteria:

1. The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic therapy (cytokines, antibodies) within 3 weeks (or nitrosoureas or mitomycin C within 6 weeks) before the first dose of XL888.
2. The subject has received prior treatment with a small molecule kinase inhibitor (including an investigational kinase inhibitor) or hormonal therapy within 14 days before the first dose of XL888.
3. The subject has received any other type of investigational agent within 28 days before the first dose of study treatment.
4. The subject has a previously-identified allergy or hypersensitivity to components of the study treatment formulation.
5. The subject has not recovered from clinically-meaningful toxicity due to prior therapy.
6. The subject has been previously treated with an HSP90 inhibitor
7. The subject has untreated or uncontrolled brain metastases or evidence of leptomeningeal involvement of disease.
8. The subject is currently receiving anticoagulation with therapeutic dose of warfarin.
9. The subject has uncontrolled intercurrent illness including, but not limited to: ongoing or active infection; diabetes mellitus; hypertension; symptomatic congestive heart failure, unstable angina pectoris, stroke or myocardial infarction within 3 months.
10. The subject has a baseline corrected QT interval (QTc) > 460 ms.
11. The subject is pregnant or breastfeeding.
12. The subject is known to be positive for the human immunodeficiency virus (HIV).
13. The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose of oral administration of XL888 when administered on an intermittent schedule to adults with solid tumors | Assessed at several visits during weeks 1 through 4 of the first cycle and approximately every other week each cycle thereafter
Plasma pharmacokinetics of oral administration of XL888 when administered on an intermittent schedule | Assessed at several visits during weeks 1 through 4 of the first cycle and approximately once every four weeks each cycle thereafter

SECONDARY OUTCOMES:
Pharmacodynamic effects of XL888 on both tumor tissue and non-tumor tissue | Assessed at specific visits during the first cycle; mandatory blood samples collected once every four weeks every cycle thereafter with optional tissue samples
Estimate renal elimination of XL888 | Assessed during the first cycle after three weeks of dosing
Exploratory: To evaluate preliminary antitumor activity of XL888 | Assessed every eight weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas